CLINICAL TRIAL: NCT01322373
Title: Improved Diagnosis of Alzheimer's Disease Using Magnetoencephalography (MEG) and the Synchronous Neural Interaction™ Test: A Follow-up Study
Brief Title: A Study of Alzheimer's Disease Using Magnetoencephalography (MEG) and the Synchronous Neural Interaction™ Test
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Orasi Medical, Inc. (Industry)
Responsible Party: Todd Verdoorn, PhD, Chief Scientific Officer, Orasi Medical, Inc.
Other Study IDs: ADG 11-01
Record Dates: First submitted 2011-03-22; First posted 2011-03-24 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2011-03

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; magnetoencephalography; MEG; SNI
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy control subjects (HC): Subjects who met criteria as healthy control subjects and completed Orasi Protocol ADG-08-01.
- Alzheimer's disease subjects (AD): Subjects with a diagnosis of DAT according to DSM-IV-TR criteria who completed Orasi Protocol ADG-08-01.

SUMMARY:
This follow-up study is designed to obtain longitudinal clinical and MEG scan data to gain information on Alzheimer's disease (AD) progression, the stability of healthy control (HC) MEG scan data, to enrich the Orasi database of AD and HC subjects, and is intended to extend the capabilities of the Synchronous Neural Interaction® (SNI) test, which is under development by the sponsor, Orasi Medical. The current study is intended to extend the database of AD and HC MEG scans and will include patients who previously enrolled and completed Orasi Protocol ADG 08-01. This study will include MEG scans on up to approximately 50 AD subjects and 70 HC subjects. Additionally, AD subjects will complete 3 standard functional tests while HC subjects will complete 2 standard functional tests. ApoE genotyping also will be determined for all subjects. The results generated in this study will be used to improve the accuracy of the SNI test for diagnosing and tracking the progression of AD.

ELIGIBILITY:
Inclusion Criteria:

* Subject enrolled and completed Orasi Protocol ADG 08-01
* Subject understands the study procedures and agrees to participate in the study by giving written informed consent. In the event the subject lacks the capacity to sign the consent form then the subject's Legally Authorized Representative (LAR) may sign on the subject's behalf. See Section 5. Informed Consent for details.
* Subject is a non-smoker.
* Subject is judged to be in good health other than AD, if applicable

Exclusion Criteria:

* Subject has a history or diagnosis of a significant neurological condition other than Alzheimer's disease including Parkinson's disease, vascular dementia, Lewy body dementia, frontal temporal dementia, human immunodeficiency virus, multiple sclerosis, seizures, epilepsy, stroke, ADHD, dyslexia, or severe traumatic brain injury.
* Subject has a history of primary psychotic disorder (e.g. schizophrenia, schizoaffective disorder, delusional disorder) or bipolar disorder.
* Subject has a Modified Hachinski Ischemia Scale (HIS) score greater than 4.
* The subject has a recent history (within 2 years) of alcohol or substance abuse/dependence.
* Subject had an MRI within two weeks prior to Study Visit 2.
* Subject has metal dental braces, pacemaker or other common medical devices that may interfere with the MEG scan.
* Subject is unable to complete the MEG scan procedure.
* Investigator has any concern regarding the safe participation of a subject in the study, or if for any other reason the investigator considers the subject inappropriate for study participation

Ages: 20 Years to 92 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects who enrolled and completed Orasi Protocol ADG 08-01 will be contacted and invited to participate in this follow-up study.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Identification and characterization of patterns of correlated brain activity measured by MEG and the Orasi SNI test that differ consistently between HC and AD subjects. | Up to 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Richard Golden, MD, Principal Investigator — Noran Neurological Clinic
Locations (2):
- United States (2):
  - Noran Neurological Clinic, Minneapolis, Minnesota
  - Noran Neurology Clinic, Plymouth, Minnesota